CLINICAL TRIAL: NCT05065996
Title: Prediction of Aortic Dilation and Rupture in Different Predisposing Pathologies A Prospective Clinical Study
Brief Title: Prediction of Aortic Dilatation and Rupture
Acronym: DilAo
Status: Completed | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other); JAMK University Of Applied Sciences (Other)
Responsible Party: Principal Investigator, Marja Hedman, Professor, Kuopio University Hospital
Other Study IDs: 5063566
Record Dates: First submitted 2021-09-14; First posted 2021-10-04 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Aortic Rupture
Keywords: aortic dilatation; aortic aneurysm; 4D flow MRI; aortic rupture
MeSH Terms: conditions — Aortic Rupture; Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Different 4D flow MRI parameters in aortic dilatation and controls: Patients with aortic dilatation (n=20) scheduled for aortic MRI and healthy controls (n=20) without aortic dilatation. One time aortic MRI with 4D flow imaging.
  Interventions: Diagnostic Test: Aortic MRI + 4D flow MRI
- Value of aortic 4D flow MRI parameters to predict aortic dilatation in 5 years follow up: Patients with aortic dilatation (n=100) scheduled for aortic MRI follow up in Kuopio University Hospital. Aortic 4D flow MRI will be done yearly for 5 years and flow parameters predicting aortic dilatation will be analysed.
  Interventions: Diagnostic Test: Aortic MRI + 4D flow MRI
- Histology, molecular biology and genetics behind aortic dilatation: Patients scheduled for aortic operation (n=20+100) in Kuopio University Hospital. Aortic tissue samples and blood will be collected for analysis and compared to 4D flow MRI parameters. Control samples will be collected from healthy organ donors (n=5+5) operated in Kuopio University Hospital.
  Interventions: Diagnostic Test: Aortic MRI + 4D flow MRI

INTERVENTIONS:
Diagnostic Test: Aortic MRI + 4D flow MRI — Together with routine aortic MRI specific 4D flow MRI sequence will be done.

SUMMARY:
Aortic aneurysm is a very common incidental finding in the diagnostic imaging of the chest. It is especially common in middle aged men (up to 40 %). It is called as a silent killer, since it can lead to aortic dissection and rupture without pre-existing symptoms. Mortality of rupture can be up to 50 %. This is why it causes extensive human uncertainty and fear. Currently, there are no methods to identify the high risk patients. That leads to a practice where all patients are followed with repeated aortic imaging using expensive methods such as magnetic resonance imaging (MRI) and computed tomography.

There is data, that modern 4D flow MRI parameters well describe the intra-aortic flow conditions. This prospective clinical trial explore the value of 4D flow MRI parameters in the prediction of aortic dilatation and rupture. The trial consists of three subtrials in whitch the 4D flow MRI parameters are tested in clinical practice.

DETAILED DESCRIPTION:
1. Purpose of the study The purpose of this study is to explore prognostic parameters for aortic dilation. More specifically it is to identify prognostic imaging parameters which could be used to identify patients at high risk for rapid aortic dilation and should be intensively followed by imaging methods.

2. Subtrials

1. Clinical study 1 The aim of the first phase of the study targets to identify 4D MRI flow parameters which are characteristic to dilated aorta and might be used to evaluate future prognosis in patients with aortic dilatation or predisposing factors.
2. Clinical study 2 The second phase of the study aims to use identified flow parameters in clinical imaging follow up to find out which parameters predict aortic dilation in real life and thus could be used to select patients for more intensive imaging in future.
3. Study 3 - Molecular pathology, histology and genetics of aorta The aim of this part of the study is to find out differences in molecular biology, histology, elasticity and genetics of the aorta in patients having predisposing factors for aortic dilation. Particularly, cellular factors influencing the formation of connective tissue and vascular smooth muscle layer will be studied.

3. Methods

1. Patient population All patients and healthy volunteers will give their written informed consent for the study. The Ethical Committee of Northern Savo hospital district has given approval for the trial.

Study 1 The first phase of the study will include twenty patients with anatomical or functional BAV or other disease predisposing to dilation of aorta scheduled for routine aortic MRI in Kuopio University Hospital (KUH) Department of Radiology. 4D flow MRI will be done right after the routine 2D MRI and it will extend the imaging time approximately 20 minutes. Twenty healthy voluntary controls will be recruited from the research group and personnel of the department and they will be scheduled for the similar imaging procedure. The main parameters analyzed from this one-off imaging data are peak flow velocity and eccentricity of the flow, flow vorticity and wall shear stress. Also, parameters related to aortic stiffness and geometry will be determined in this study. Comparison of the 4D flow MRI parameters between the patients and healthy controls will be done, 4D flow parameters will also be compared to conventional 2D flow parameters both in the study patients and in healthy controls.

Study 2 For the follow-up study 100 patients will be recruited on the same manner as in the case of the first study patients. The inclusion criteria will be: adult (age > 18 years), previously documented aortic dilation, documented anatomical or functional BAV or other inherited disorder, which caus-es increased risk for aortic dilation, no contraindication for MRI. Similar aortic MRI will be performed as during the clinical study 1. However, the follow-up imaging will be performed after 6 months from the first MRI and yearly for 5 years. Same 4D and 2D flow parameters will be analyzed as in the first study. The special interest will be appointed to the degree of aortic dilation and correlation between 4D (and 2D) flow parameters to the aortic dimensions.

Clinical parameters All patients visiting outpatient clinic will have clinical examination (auscultation, clinical signs for heart failure, hepatomegaly, peripheral edema, arterial murmurs). 12-lead electrocardiography and basic laboratory analyses (hemoglobin, hematocrit, sodium, potassium, creatinine, brain natriuretic peptide) will be performed. With patient written permission, an additional tube of blood will be saved for future analysis and the patient will be informed about the purpose of this sample.

Echocardiography Transthoracal echocardiography will be done by using routine clinical methods. Special interest will be appointed to aortic valve anatomy and aortic dimensions. Other signs of cardiac mani-festations will also be registered. Ventricular dimensions and volumetric parameters as well as ventricular systolic and diastolic function will be evaluated.

Aorta MRI Magnetic resonance angiography and 2D flow measurements Static imaging of the aorta is done with an ECG- and respiratory-gated 3D SSFP (steady state free percession) sequence [Kawel et al 2012]. Image stack is obtained in sagittal plane and processed at the MPR-workstation to get images perpendicular to the axis of blood flow. The diameter of the aorta is measured from outer wall to the outer wall. The widest diameter of the aorta is de-termined and, as a routine, diameter of the aorta is measure at 8 pre-determined levels.

4D phase contrast MRI Blood flow in the aorta will be measured based on MRI phase contrast. The measurement will be done by repeating the imaging pulse sequence without and with flow weighting gradients for three dimensions with interleaved manner and the measurement. The imaging parameters will be set according to 4D MRI flow measurement consensus statement [Dyverfelt 2015] shortly: resolution of < 2.5x2.5x2.5 mm3, temporal resolution of 30 ms (time resolution in flow in different cardiac phases), retrospective ECG synchronization and respiratory motion compensation, flip an-gle close to Ernst angle and the flow weighting gradient amplitude so that maximum flow of 10 % higher than expected maximum flow rate in the aorta. The imaging volume will be cover the aor-tic valve, aortic arc and descending aorta at the level of apex of myocardium. The data will be preprocessed to minimize contribution from background phase offsets, gradient imperfections and phase wraps.

Flow parameters From the 4D flow images, several quantitative parameters will be extracted. The main parame-ters are the ones describing flow distribution in the aorta, i.e. peak flow velocity and eccentricity, flow vorticity and shear stress on the vessel walls. Furthermore, several parameters related to aortic stiffness and geometry and function of aortic valve, will be recorded. During follow-up, changes and prognostic value of the quantified parameters will be evaluated.

In the purpose of validation 4D flow parameters will be compared to parameters extracted from conventional 2D flow sequences.

Clinical follow-up protocol Patients recruited for the follow up study (study 2) will be re-screened by aortic MRI after half year from the recruitment and yearly after the first follow-up visit up to five years or according to clinical follow-up schedule. If the state of the aortic dilation indicates more intensive follow-up will be used.

Statistical analyses Prognostic factors will be tested for statistical significance by comparing flow parameters and as-sociated factors to the degree of aortic dilation by using appropriate multivariate analysis . Statis-tical significance will be set at p<0.05 and high statistical significance at p < 0.01. The data will be analyzed by using SPSS for Windows program.

Study 3

The third subtrial will enroll 20+100 patients with severe aortic dilatation scheduled for aortic operation. Human aorta samples are collected during routine aorta replacement surgery from the removed vascular tissue. In addition to tissue samples, a blood sample will be collected for genetic and molecular analysis. Patients have given their written permission for the histological and blood samples before the operation. After resection, samples are immediately transferred into liquid nitrogen (frozen samples), PFA-PBS (histological samples) or to cell culture medium for cell isolation (endothelial cells, vascular smooth muscle cells, fibroblasts). Frozen samples are stored in -70 °C and isolated cells in liquid nitrogen. Histological samples will be processed into the paraffin and stored as a paraffin blocks. Samples will be stored up to 10 years, and after which they are destroyed as a biohazard waste. Raw data will be stored in electrical archive like European Genome-phenome Archive (EGA).

Analyses Molecular biology and histology of the aorta samples are examined by RT-qPCR, immunohisto-chemistry and multiphoton microscopy imaging. Expression of relevant genes e.g. TGF-β, VEGF-family, COX-1 and 2, eNOS/Akt and pro-inflammatory cytokines is studied, and also RNA -sequencing, identifying all expressed mRNAs simultaneously, can be used for finding differences in expression of all aortic genes between different patient groups. FBN1 gene is sequenced and looked for mutations or deletions.

Aorta vessel wall architecture and expression of relevant genes is visualized by multiphoton mi-croscopy and immunohistochemistry. Isolated cells are used for Single Cell Analysis, which allows studying one living cell and its molecular events at a time, and gives totally new information about functions of different cells in vessel wall. Obtained data is divided in disease- and age matching groups, and correlations between cardiac disease status, aortic gene expression and aortic histology will be looked for. Data will also be connected and compared to the pre-clinical mouse study described in Appendix 1, and human aorta MRI 4D flow imaging study described in paragraph 3.4.

Biomechanics of histological aorta samples Biomechanical parameters such as the stiffness and failure strength will be measured from the aorta samples. The measurements and analysis will be done in collaboration with The BBC group in University of Eastern Finland. The biomechanical parameters in the studied patients groups will be compared and used as a parameter in multivariant statistical analyses. The results will also be compared and linked to findings of histological and molecular biology.

Controls Samples for comparison to normal tissue will be collected from 10 organ donors operated in Kuopio University Hospital. The samples will be handled as described in aortic patients.

Mathematic modelling of aorta Imaging data of 20 patients will be send anonymously to JAMK University of Applied sciences for mathematic simulation modelling of aortic flow and wall stress.

4. Collaboration The clinical study is conducted multiprofessionally in Kuopio University Hospital together with departments of clinical cardiology, cardiothoracic surgery (Heart Center) and radiology (Clinical Imaging Center). The histopathological, molecular and genetic studies are performed in the Department of Molecular Sciences in A I Virtanen Institute, University of Eastern Finland (UEF). Biomechanical tests will be conduited in the Department of Applied Physics in UEF.The mathematic modelling of the aortic images will be performed in JAMK University of Applied Sciences. The acquired 4D MRI flow results will be analyzed and validated according to standards of Kuopio University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* aortic dilatation
* scheduled for imaging follow up in Kuopio University Hospital
* written informed concent

Exclusion Criteria:

* lack of co-operation
* contraindications to MRI

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Patients with aortic dilatation scheduled for follow up in Kuopio University Hospital
  * Patients with aortic dilatation scheduled for aortic operation in Kuopio University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Association of WSS to aortic dilatation rate | 5 years
  4D flow MRI wall shear stress value in correlation to aortic diameter in different time points
Association of FD to aortic dilatation rate | 5 years
  4D flow MRI flow displacement value in correlation to aortic diameter in different time points

OTHER OUTCOMES:
Association of WSS and FD to histology | 2 years
  hematoxylin eosin, CD31, inflammatory cells of human aortic samples in correlation to WSS and FD
Association of WSS and FD to genetics | 2 years
  Gene screening from human blood samples of aortic patients

CONTACTS AND LOCATIONS:
Overall Officials: Marja Hedman, Prof, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No
only anonymous imaging data will be send to JAMK university of applied sciences for mathematical modelling of aorta

REFERENCES:
- [Derived] Kiljander T, Kauhanen P, Sillanmaki S, Lottonen-Raikaslehto L, Husso M, Yla-Herttuala E, Saari P, Kokkonen J, Laukkanen J, Mustonen P, Hedman M. Repaired coarctation of the aorta does not affect four-dimensional flow metrics in bicuspid aortic valve disease. Interdiscip Cardiovasc Thorac Surg. 2024 May 2;38(5):ivae086. doi: 10.1093/icvts/ivae086. PMID 38704861